CLINICAL TRIAL: NCT03202277
Title: BeWell24: Smartphone-based Diabetes Prevention in the VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R18DK109516 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: physical activity, sleep, sedentary behavior, dietary intake, smartphone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeWell24 smartphone app (Experimental): Smartphone app, linked with commercial activity monitor, to support lifestyle changes in physical activity, sleep, sedentary behavior, and dietary intake.
  Interventions: Behavioral: BeWell24 smartphone app
- Health education smartphone app (Active Comparator): Smartphone app with basic health education content, designed to control for non-specific treatment effects and match for smartphone app novelty.
  Interventions: Behavioral: Health education app

INTERVENTIONS:
Behavioral: BeWell24 smartphone app — This app delivers an evidence-based suite of lifestyle interventions targeting behavior change in sleep, sedentary behavior, physical activity, and dietary intake. The app connects with a commercially available activity monitor to provide real-time feedback on behaviors over time.
  Arms: BeWell24 smartphone app
Behavioral: Health education app — This app delivers basic health education and hygiene content related to sleep, sedentary behavior, physical activity, and dietary intake.
  Arms: Health education smartphone app

SUMMARY:
Type 2 diabetes (T2D) is a national epidemic and current lifestyle programs and medications are not effectively managing the crisis. This project aims to test a novel smartphone-delivered intervention that simultaneously targets multiple health behaviors (i.e., sleep, sedentary behavior, physical activity,dietary intake) within clinical settings at a large Veteran Health Administration regional hospital. If effective, this project has potential for large-scale implementation nationwide through the VA healthcare system and broad applicability for other populations at T2D risk as well as other disorders.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) affects 26 million Americans and "prediabetes" affects 86 million more. If this epidemic is not addressed immediately, 23% of Americans will have T2D by 2030. Current lifestyle programs to prevent diabetes are complex to deliver, costly, and have limited scalability. Medications do not clearly modify the disease process and have a number of side effects. New approaches are needed that can address this epidemic on a population scale. mHealth technologies (e.g., smartphones) are deeply integrated into our lives and can target the daily lifestyle behaviors that underpin the T2D epidemic. The Veterans Health Administration (VHA) is an ideal setting to test mHealth approaches because they are at the forefront of harnessing smartphone technologies to deliver care with the advent of the "VA App Store." As the nation's largest integrated healthcare system, VHA has a central dissemination infrastructure to deliver smartphone interventions to over 5.5 million Veterans. BeWell24, an adaptive and multicomponent smartphone "app" was developed based on the unique needs and desires of US Veterans and VHA clinical teams. BeWell24 targets behaviors across the 24 hours - sleep, sedentary behavior, and more active behaviors - and preliminary data suggest reductions in fasting glucose among prediabetics of 12.3% in just 8 weeks of use. A dietary component will be added to the app to further enhance the potency of the intervention. The objective now is to test whether the delivery and integration of this app into routine clinical care settings can improve glycemic control over 9 months. A randomized controlled trial of 120 prediabetic Veterans is proposed. The first aim is to test whether BeWell24 significantly improves glycemic control (reduce fasting glucose and HbA1c) over 9 months relative to usual care. Objectively-measured changes is targeted behaviors (sleep, sedentary behavior, physical activity, and dietary intake) and other key cardiometabolic biomarkers (weight/body fat, blood pressure, lipids, insulin, and hs-CRP) will also be explored. The second and third aims are to assess factors impacting scalability of BeWell24 from patient and provider perspectives to optimize opportunities for large-scale dissemination if efficacious. Program reach/retention, app usage, treatment acceptability, program costs, and clinical integration factors will be studied. Unique features of this proposal are the rigorous cluster-randomized design; testing in a highly integrated, nationwide, clinical setting; and use of a highly sophisticated smartphone platform uniquely designed for the population and targets multiple health behaviors impacting T2D risk. The long-term goal is to establish an effective diabetes prevention program among Veterans that can be used to complement and enhance existing clinical support. If effective, this approach could be rapidly scaled to Veterans nationwide and could have broad applicability for other populations at disparate T2D risk as well as other disorders.

ELIGIBILITY:
Inclusion Criteria:

* Veterans ages 18 and older
* Regularly use an appropriate Apple (iOS6 or higher) or Android (2.3 or higher) smartphone or tablet device
* Risk for "prediabetes" based upon clinician judgment - clinicians may rely on laboratory data review in the prior 12 months including: (a) HbA1c 5.7-6.4%; and (b) glucose, HDL-cholesterol, triglycerides, and weight

Exclusion Criteria:

* long distance or insufficient transportation to the Veterans hospital to make participation in quarterly visits difficult;
* severe personal, health, cognitive or psychological conditions that prevent participation or severely limit lifestyle changes
* limited physical mobility, untreated sleep disorder, or other underlying disorder that requires treatment or would make lifestyle change contraindicated
* current participation in other diet, weight loss, or lifestyle programs
* recent or imminent changes in medications that would substantially alter glucose metabolism (e.g., steroids, anti-depressive medications associated with weight gain)
* recent weight gain or loss of more than 10 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
HbA1c | 9 months
  Circulating levels of Hemoglobin A1c
Fasting glucose | 9 months
  Fasting levels of glucose

SECONDARY OUTCOMES:
Sleep duration (minutes/night) measured by wrist actigraphy | 9 months
  Sleep duration (measured by wrist actigraphy)
Sedentary behavior (minutes/day) measured by wrist actigraphy | 9 months
  Measure of sedentary time (measured by wrist actigraphy)
Moderate-vigorous physical activity (minutes/day) measured by wrist actigraphy | 9 months
  Measure of moderate-vigorous physical activity (measured by wrist actigraphy)
Dietary quality measured by the NCI dietary factor screener | 9 months
  Self-reported dietary quality

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - Arizona State University, Tempe, Arizona

IPD SHARING:
Plan to Share IPD: No